CLINICAL TRIAL: NCT04439448
Title: An Observational Cohort Study of Adipose Tissue and Immune Activation in Treated HIV Infection
Brief Title: Adipose Tissue and Immune Activation in HIV
Acronym: AIAC
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, John R. Koethe, Associate Professor, Vanderbilt University Medical Center
Other Study IDs: K23AI100700 (NIH)
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Human Immunodeficiency Virus; Obesity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Obesity | interventions — Absorptiometry, Photon; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV+ non-obese: HIV+ adults on antiretroviral therapy with a body mass index <30 kg/m2
  Interventions: Radiation: dual-energy X-ray absorptiometry (DEXA) scan; Other: Carotid and branchial artery ultrasound; Diagnostic Test: 2-hour oral glucose tolerace test; Diagnostic Test: Blood collection
- HIV+ obese: HIV+ adults on antiretroviral therapy with a body mass index >=30 kg/m2
  Interventions: Radiation: dual-energy X-ray absorptiometry (DEXA) scan; Other: Carotid and branchial artery ultrasound; Diagnostic Test: 2-hour oral glucose tolerace test; Diagnostic Test: Blood collection
- HIV-negative obese: HIV-negative adults on antiretroviral therapy with a body mass index >=30 kg/m2
  Interventions: Radiation: dual-energy X-ray absorptiometry (DEXA) scan; Other: Carotid and branchial artery ultrasound; Diagnostic Test: 2-hour oral glucose tolerace test; Diagnostic Test: Blood collection

INTERVENTIONS:
Radiation: dual-energy X-ray absorptiometry (DEXA) scan — Whole body dual-energy X-ray absorptiometry (DEXA) scan to assess lean and fat mass
Other: Carotid and branchial artery ultrasound — Ultrasound to assess carotid plaque and brachial artery flow mediated dilation
Diagnostic Test: 2-hour oral glucose tolerace test — Ingestion of 75g of glucose syrup with blood collection for glucose and insulin at time 0, 90min and 120min
Diagnostic Test: Blood collection — Blood collection for measurement of circulating proteins (cytokines) and isolation of immune cells

SUMMARY:
The prevalence of HIV-associated wasting declined dramatically with the introduction of effective antiretroviral therapy (ART), but as patients survive longer on treatment the proportion of overweight (body mass index [BMI] >25 kg/m2) and obese (BMI >30 kg/m2) HIV-infected individuals has been rising over time and is reaching parity with the general population. Adipose tissue has broad effects on immune function relevant to HIV infection, including the basal inflammatory state and peripheral lymphocyte populations, but there are few data on the effects of high adiposity on HIV immunology. This issue is directly relevant to promoting the long-term health of ART-treated individuals, many of which can now survive for decades on treatment, as emerging evidence suggests that increased immune activation is a major risk factor for the development of cardiovascular and metabolic diseases in this population. HIV-infected individuals on ART have an approximately 2-fold higher risk of myocardial infarction and a 4-fold higher risk of type 2 diabetes mellitus, and the proportion of deaths among HIV-infected individuals due to non-AIDS conditions now exceeds those due to AIDS.

Despite the increasing proportion of overweight and obese HIV-infected persons, few prior studies have investigated the interaction between adipose tissue, immune activation, and risk factors for cardiovascular and metabolic disease in treated HIV. The overall goal of this study is to understand the complex relationships between adipose tissue, innate and cellular immune activation, and metabolic and cardiovascular disease risk factors in persons on long-term antiretroviral therapy. To this end, we will use an observational, cross-sectional cohort design to compare in vivo markers of immune activation, ex vivo cytokine expression, and metabolic and cardiovascular disease markers in HIV-infected individuals with a range of body composition profiles and between overweight/obese HIV-infected and uninfected individuals.

DETAILED DESCRIPTION:
HIV-infected individuals on long-term ART treatment are at increased risk for many diseases, particularly diabetes mellitus and coronary artery disease, which are more commonly associated with obesity and a sedentary lifestyle. As HIV patients are now living longer on effective treatment, a growing proportion are becoming overweight and obese, and the management of non-AIDS chronic diseases associated is emerging as a major challenge to clinicians and the health care system. Excess adiposity (i.e., being overweight or obese) and treated HIV infection are associated with strikingly similar alterations in inflammatory biomarkers and cellular immune function implicated in the pathogenesis of chronic diseases, but there are few data at present on whether the effects of obesity and treated HIV are synergistic or additive. In this study we will closely investigate the effects of adipose tissue on both the innate and cellular arms of the immune system, and the relationships between adiposity, immune function, and risk factors for metabolic and cardiovascular diseases.

Heightened, chronic systemic inflammation is an important contributor to non-AIDS related morbidity and mortality among patients on ART, and treated HIV and obesity may promote increased metabolic and cardiovascular disease through similar mechanisms. Elevated serum highly-sensitive C-reactive protein (hsCRP; a more sensitive serum CRP assay used to measure inflammation), interleukin-6 (IL-6), and other innate immune-derived inflammatory markers are independently associated with increased risk of cardiovascular events, insulin resistance, and all-cause death among HIV-infected individuals. The etiology of this HIV-associated inflammation is not fully understood and likely multifactorial, but serum hsCRP and several proinflammatory cytokines (e.g., IL-6, TNF-α receptor 1) correlate with fat mass in HIV-infected adults, suggesting adipose tissue may have a role in modulating the inflammatory response.

In addition to greater inflammation, abdominal obesity is associated with altered T cell function, characterized by increased circulating markers of cellular immune activation (e.g., sCD25 and neopterin), and adipose tissue biopsies from obese individuals and animal models contain higher numbers of resident macrophages, T cells (particularly CD8+ cells) and reduced T-regulatory cells. Furthermore, adipokines (hormones produced by adipocytes), demonstrate a range of lymphocyte effects. Leptin, in particular, enhances expression of T cell activation markers after PHA stimulation, polarizes naïve CD4+ T cell proliferation towards the Th1 phenotype, and promotes Th1 cytokine production. These in vitro data are consistent with obesity modulating T cell activation, at least in part through adipokine effects.

The goal of this study is to understand the complex relationships between adipose tissue, innate and cellular immune activation, and metabolic and cardiovascular disease risk factors in persons on long-term antiretroviral therapy. Using the facilities and resources of the Vanderbilt Clinical Research Center, we will enroll an observational cohort to investigate the interactions of innate immune activation, metabolic and cardiovascular risk factors, and T cell activation among HIV-infected and uninfected adults with a range of body composition profiles from low adiposity (lean) to high adiposity (obese). The study groups will be comprised of 70 HIV-infected adults on ART with a range of body composition profiles from low adiposity (lean) to high adiposity (obese), and a control group of 30 overweight and obese uninfected individuals.

Hypothesis 1: Increased adipose tissue promotes increased innate and cellular immune activation in HIV-infected individuals on long-term ART.

Specific Aim 1a: To study the hypothesis that adipose tissue promotes innate immune activation in treated HIV by determining if serum leptin (a marker of adiposity) is positively associated with interleukin-6 (IL-6) levels, in addition to other inflammation biomarkers (including C-reactive protein), in HIV-infected persons on long-term ART with a range of body composition profiles from low adiposity (lean) to high adiposity (obese).

Specific Aim 1b: To study the hypothesis that adipose tissue promotes cellular immune activation in treated HIV by determining if serum leptin is positively associated with the percentage of CD8+ T cells expressing CD38 and HLA-DR activation markers in HIV-infected persons on long-term ART.

Hypothesis 2: Overweight and obese HIV-infected individuals on long-term ART have significantly greater markers of innate and cellular immune activation compared to uninfected individuals with equivalent adiposity.

Specific Aim 2a: To determine if IL-6 serum levels, and other inflammation biomarkers, are significantly higher among overweight/obese HIV-infected persons compared to uninfected controls with equivalent adiposity.

Specific Aim 2b: To determine if the percentage of CD38+ and HLA-DR+ CD8+ T cells is significantly higher among overweight/obese HIV-infected persons compared to uninfected controls with equivalent adiposity.

ELIGIBILITY:
HIV-infected participants:

Inclusion Criteria:

* age >18 years
* on ART >2 years
* a CD4+ nadir >100 cells/µl prior to starting ART
* a CD4 >350 cells/µl at the time of enrollment
* HIV-1 viral load <50 copies/ml
* Pre-menopausal

Exclusion Criteria:

* Pregnant (women only)
* Current use of anti-diabetic medications or statins

HIV uninfected participants:

Inclusion Criteria:

* age >18 years
* body mass index >= 30 kg/m2
* Pre-menopausal

Exclusion Criteria:

* Pregnant (women only)
* Current use of anti-diabetic medications or statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health persons with HIV receiving care at the Vanderbilt Comprehensive Care Clinic and healthy persons without HIV receiving care at Vanderbilt University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-04-12 (Actual); Primary Completion 2014-11-03 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
CD38+ CD4+ T cells | At study enrollment
  Flow cytometry measurement of CD38 expression on isolated CD4+ T cells
Plasma interleukin-6 | At study enrollment
  Level of circulating interleukin-6

SECONDARY OUTCOMES:
Carotid intima media thickness | At study enrollment
  Ultrasound measurement of carotid intima media thickness
Brachial artery maximal flow mediated dilation | At study enrollment
  Ultrasound measurement of maximal brachial artery dilation after 5 minutes of hypoxia
Visceral adipose tissue volume (cm3) | At study enrollment
  Dual-energy x-ray assessment of visceral adipose tissue volume

CONTACTS AND LOCATIONS:
Overall Officials: John Koethe, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time to share IPD with other researchers. There have been no requests to share data.

REFERENCES:
- [Result] Koethe JR, Jenkins CA, Furch BD, Lake JE, Barnett L, Hager CC, Smith R, Hulgan T, Shepherd BE, Kalams SA. Brief Report: Circulating Markers of Immunologic Activity Reflect Adiposity in Persons With HIV on Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):135-140. doi: 10.1097/QAI.0000000000001768. PMID 29794823
- [Result] Grome HN, Barnett L, Hagar CC, Harrison DG, Kalams SA, Koethe JR. Association of T Cell and Macrophage Activation with Arterial Vascular Health in HIV. AIDS Res Hum Retroviruses. 2017 Feb;33(2):181-186. doi: 10.1089/AID.2016.0113. Epub 2016 Sep 14. PMID 27527002
- [Result] Koethe JR, Jenkins CA, Petucci C, Culver J, Shepherd BE, Sterling TR. Superior Glucose Tolerance and Metabolomic Profiles, Independent of Adiposity, in HIV-Infected Women Compared With Men on Antiretroviral Therapy. Medicine (Baltimore). 2016 May;95(19):e3634. doi: 10.1097/MD.0000000000003634. PMID 27175676
- [Result] Koethe JR, Grome H, Jenkins CA, Kalams SA, Sterling TR. The metabolic and cardiovascular consequences of obesity in persons with HIV on long-term antiretroviral therapy. AIDS. 2016 Jan 2;30(1):83-91. doi: 10.1097/QAD.0000000000000893. PMID 26418084
- [Result] Masenga SK, Elijovich F, Hamooya BM, Nzala S, Kwenda G, Heimburger DC, Mutale W, Munsaka SM, Zhao S, Koethe JR, Kirabo A. Elevated Eosinophils as a Feature of Inflammation Associated With Hypertension in Virally Suppressed People Living With HIV. J Am Heart Assoc. 2020 Feb 18;9(4):e011450. doi: 10.1161/JAHA.118.011450. Epub 2020 Feb 17. PMID 32064996